CLINICAL TRIAL: NCT04704674
Title: Community Dynamics of Malaria Transmission in Humans and Mosquitoes in Fleh-la and Marshansue, Salala District, Bong County, Liberia
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000158; 000158-I
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01-06

CONDITIONS: Malaria
Keywords: Assays; BLOOD SAMPLING; Parasites; Gametocyte; Infection; Natural History
MeSH Terms: conditions — Malaria; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 0.5 - 5 years: Age bracket for infants/children up to age five years
- 10 - 18 years: Age bracket for children 10 - 18 years
- 19 + years: Age bracket for adults over 19 years
- 5 - 10 years: Age bracket for children ages 5 - 10 years

SUMMARY:
Background:

Malaria is a disease that affects many people in Liberia. It is caused by germs (parasites) that are spread by mosquito bites. Researchers want to gather data that may help them understand the best way to use a malaria vaccine in Liberia, which will be important in getting rid of the disease.

Objective:

To find out how often people of all ages who live in Fleh-la and Marshansue, Liberia, get malaria.

Eligibility:

Healthy people ages 6 months and older who live in Fleh-la and Marshansue in a household with adults and children.

Design:

Participants will be screened with a physical exam and questions about their health.

Participants will have monthly study visits. They will be asked about any symptoms of malaria and their use of bednets. Their vital signs, such as blood pressure and temperature, will be checked. Blood will be taken from the participant s arm or finger with a needle. If they have a fever, they will get a malaria test. If positive, they will get drugs to treat malaria.

Once a month, participants houses will be examined for mosquitoes. The team will remove all mosquitoes they collect. As part of this collection, participants houses will be sprayed with a chemical to kill mosquitoes and other insects. Participants will not be allowed in their house while the team is inside. The spray will not harm the participants.

Once a year, at the monthly visit, an additional blood sample will be taken.

Some of the participants blood samples will be used for genetic testing.

Participation will last for up to 3 years.

DETAILED DESCRIPTION:
A vaccine that interrupts malaria transmission is critical to eradicate the disease, but improved assays are needed to measure the efficacy of vaccines. Transmission-blocking vaccines (TBVs) work by inducing antibodies that inhibit parasite development in the mosquito interrupting transmission. Efficacy of vaccines may be estimated by in vitro membrane feeding assays using immune sera and laboratory mosquitoes, but qualified assays that measure transmission in the field are needed to assess transmission-blocking interventions in natura. Clinical trials of TBVs have started elsewhere on the continent in Mali, and we have planned to expand TBV studies here in Liberia soon. This protocol is already being used for a longitudinal cohort to gather information of malaria transmission based on the rates of blood smear positive individuals by month, season and year in Fleh-la and Marshansue, in Salala, Bong County, Liberia. Individuals in the villages were approached first for participation, including permission to contact their household and neighbors of their compound for participation. Households were identified using census data and individuals who consented for participation are being enrolled. Malaria smears are obtained at monthly visits, in conjunction with mosquito collections in/around village residences. Parasite infection rates in locally caught mosquitoes will be assessed longitudinally for differences by season and year. A total of 400 volunteers from Fleh-la and Marshansue will be enrolled. Participants will be followed for at least one year, to collect data that will guide the design of future community-based trials of TBV for which this amendment is being submitted for approval.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject Inclusion Criteria:

* 6 months of age and above
* Known resident of Fleh-la and Marshansue or the surrounding villages and planning to remain for duration of study
* Willingness to allow stored laboratory specimens to be used for future research
* Acceptance and signature of the written informed consent and the assent for children aged 12-17 years who are not otherwise emancipated

Household Inclusion Criteria:

To be eligible for participation, households must meet the following criteria:

* Household with at least 3 residents eligible for participation.
* Household with at least one compound member who is below 18 years of age whose parents or caretakers are willing to provide informed consent for the child to participate.
* Household members willing to accommodate mosquito sampling in their compound, both indoors and outdoors.

Exclusion Criteria:

Subject Exclusion Criteria:

* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An estimated total of 400 volunteers from Fleh-la and Marshansue and surrounding villages will be enrolled. Participants above the age of six months will be approached to participate in the study; and will be followed for up to 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Measurement of Monthly rates of blood smear positive individuals by age | one year
  Rate of blood smear positive individuals

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Hume, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Public Health Institute of Liberia (NPHIL), Fleh-la, Liberia

IPD SHARING:
Plan to Share IPD: No